CLINICAL TRIAL: NCT01608243
Title: Investigation of the Safety, Tolerability and Pharmacodynamic Effects of Sublingual Immunotherapy Tablets of House Dust Mite Allergen Extracts in Adults With House Dust Mite-associated Allergic Asthma
Brief Title: Safety Study of Sublingual Immunotherapy Tablets of House Dust Mite Allergen Extracts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO71.11
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Asthma; House Dust Mite Allergy
MeSH Terms: conditions — Asthma; Dust Mite Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLIT tablets of HDM allergen extracts (Experimental)
  Interventions: Biological: SLIT tablets of house dust mite allergen extracts
- Placebo (Placebo Comparator)
  Interventions: Biological: Matching placebo

INTERVENTIONS:
Biological: SLIT tablets of house dust mite allergen extracts — 10 dosing days
  Arms: SLIT tablets of HDM allergen extracts
Biological: Matching placebo — 10 dosing days
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety of different doses of sublingual tablets of house dust mite allergen extracts in adults with house dust mite-associated allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male or female patient from 18 to 50 years.
* Diagnosed asthma with medical history consistent with HDM-induced allergic asthma.
* Positive SPT to House Dust Mites(HDM)and HDM-specific IgE serum value ≥ 0.7 kU/L.
* Stable asthma treatments.
* Spirometry with best FEV1 > 70% of the predicted value.
* Spirometry with reversibility of FEV1 of ≥ 12% and ≥ 200 mL.
* Asthma Control Test™ (ACT) score ≥ 20.

Exclusion Criteria:

* Current smoker or former smoker with > 10 pack/year history.
* Co-sensitisation to any allergen possibly leading to clinically relevant respiratory allergy likely to significantly change the symptoms of the patient throughout the treatment period.
* Patient with a past or current disease, which as judged by the Investigator, may affect the patient's participation in or the outcome of this study.
* Patient with any oral condition that could confound the safety assessments or planning to have a dental extraction during the study.
* Female patient pregnant or breast-feeding/lactating.
* Female patient of childbearing potential not using a medically accepted contraceptive method.
* Patient treated with beta-blockers, tricyclic antidepressants or monoamine oxidase inhibitors (MAOIs).
* Patient who received allergen immunotherapy for HDM in the last 10 years.
* Ongoing treatment by immunotherapy with another allergen.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability as indicated by adverse events and safety laboratory evaluation | 10 dosing days

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Demoly, MD, Principal Investigator — CHU Arnaud de Villeneuve, Montpellier, France
Locations (1):
- CHU Arnaud de Villeneuve, Montpellier, France